CLINICAL TRIAL: NCT03403582
Title: Raspberries, Postprandial Metabolism and Type 2 Diabetes Mellitus
Brief Title: Raspberries and Postprandial Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Principal Investigator, Arpita Basu, Associate Professor, Oklahoma State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HE1465
Record Dates: First submitted 2018-01-05; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): A high-fat break fast meal with no raspberries.
- Raspberry arm (Experimental): A high-fat break fast meal with raspberries (250g frozen)
  Interventions: Other: Raspberries

INTERVENTIONS:
Other: Raspberries — 250g frozen whole red raspberries
  Arms: Raspberry arm

SUMMARY:
Raspberries are high in several phytochemicals, vitamin C and B vitamins and have been shown to be potent antioxidants and anti-inflammatory agents. However, human interventional studies reporting the effects of raspberries in obesity, T2DM and associated oxidative stress and inflammation are limited. Aims, objectives and methods:

Aim 1: To assess the effects of raspberries in postprandial glycemia and lipemia following a high-fat fast-food style meal challenge versus control group Objectives: to execute this aim, the investigators will conduct analyses of serum glucose, insulin and lipids (total cholesterol, LDL-cholesterol, triglycerides, VLDL-cholesterol and HDL-cholesterol) at fasting (baseline) and at postprandial 1,2,4 hours of high-fat, fast food style breakfast consumption. The investigators will also calculate homoeostasis model assessment of insulin resistance (HOMA-IR) at these time points using serum glucose and insulin values.

Aim 2: To assess the effects of raspberries in postprandial vascular functions (blood pressure and artery elasticity) and inflammation following a high-fat fast food style meal challenge versus control group

Objectives: to execute this aim, the investigators will measure C-reactive protein (CRP) and the following parameters of vascular function associated with CVD at fasting (baseline) and at postprandial 1,2,4 hours of high-fat, fast food style breakfast consumption:

* systolic blood pressure and diastolic blood pressure
* large artery elasticity index and small artery elasticity index
* systemic vascular resistance

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes

Exclusion Criteria:

* not having type 2 diabetes

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose | postprandial 4 hours
  Postprandial blood glucose will be measured at fasting, 1, 2 and 4 hours following meals with or without raspberries
Postprandial blood lipids | postprandial 4 hours
  Postprandial blood lipids will be measured at fasting, 1, 2 and 4 hours following meals with or without raspberries

SECONDARY OUTCOMES:
Postprandial inflammation | postprandial 4 hours
  Postprandial C-reactive protein and interleukins will be measured at fasting, 1, 2 and 4 hours following meals with or without raspberries

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No